CLINICAL TRIAL: NCT05721248
Title: The STOP-HER2 Trial: A Phase 2 Study of Stopping Trastuzumab - Outcomes in Patients With HER2+ Metastatic Breast Cancer
Brief Title: STOP-HER2: Stopping Trastuzumab in HER2+ MBC
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Gateway for Cancer Research (Other); Susan G. Komen Breast Cancer Foundation (Other); Translational Breast Cancer Research Consortium (Other); Johns Hopkins University (Other)
Responsible Party: Principal Investigator, Nancy Lin, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22-655; 1K08CA252639-01A1 (NIH)
Record Dates: First submitted 2023-02-01; First posted 2023-02-09 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Breast Cancer; Metastatic Breast Cancer; HER2-positive Breast Cancer
Keywords: Breast Cancer; Metastatic Breast Cancer; HER2-positive Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort 1: Observational Continue Anti-HER2 Therapy (No Intervention): Participants will have scans 30 days prior to starting study then undergo clinical follow-up 4-6 weeks after study initiation, at 12 weeks, and every 12 weeks thereafter. Visits will include interval history, physical exam, concomitant medications and blood draw for tumor marker assessment and research blood.
  Participants will undergo restaging scans every 12 weeks (+/- 2 weeks).
- Cohort 2: - Stop Anti-HER2 Therapy (Experimental): Participants will have scans 30 days prior to starting study. Week 1 participants will stop anti-HER2 therapy then undergo clinical follow-up every 4-6 weeks, at 12 weeks, and every 12 weeks thereafter. Visits will include interval history, physical exam, concomitant medications and blood draw for tumor marker assessment and research blood.
  Participants will undergo restaging scans every 12 weeks (+/- 2 weeks). Participants remaining progression-free after one year off treatment, may continue off anti-HER2 therapy indefinitely, with imaging surveillance suggested to be every 3-6 months at the discretion of the treating oncologist and will be followed up to 10 years Participants with disease progression after stopping anti-HER2 therapy, treatment is at discretion of the treating physician but resuming the pre-study regimen is strongly encouraged.
  Interventions: Other: Cessation of anti-HER2 treatment

INTERVENTIONS:
Other: Cessation of anti-HER2 treatment — Cessation of anti-HER2 treatment with standard treatment described as trastuzumab (Herceptin) with or without pertuzumab (Perjeta) continued as long as it is working or significant side effects occur.
  Arms: Cohort 2: - Stop Anti-HER2 Therapy

SUMMARY:
This study is being done to see if anti-HER2 treatment be safely stopped in patients with HER2-positive metastatic breast cancer (MBC) that have had exceptional response to treatment. Exceptional response" is considered as cancer progression being controlled for three years or more since starting anti-HER2 treatment.

DETAILED DESCRIPTION:
This is a single arm, phase II study of cessation of anti-HER2 systemic therapy in exceptional responders with HER2-positive metastatic breast cancer (MBC), defined as individuals free of disease progression after at least 3 years of first-line treatment.

This research study will include two different groups (cohorts) of patients. Those not wanting to stop anti-HER2 maintenance treatment will be included in a non-randomized, observational cohort (cohort 1). Those willing to stop maintenance anti-HER2 treatment you will be included in cohort 2.

This study is trying to understand whether blood samples that may contain traces of DNA from cancer, known as "circulating tumor DNA" or "ctDNA" are able to help identify which patients can successfully stop treatment without a change in their cancer.

The research study procedures include: an initial screening phase followed by periodic visits with blood work, questionnaires, and body scans.

It is expected that about 82 people will take part in this research study (52 in cohort 2 (stopping treatment), 30 in cohort 1 (continuing treatment). This study is expected to last 1 year with 10 years of follow up.

The Susan G. Komen Foundation, the Gateway for Cancer Research - both nonprofit foundations supporting cancer research - and the National Institutes of Health are supporting this research study by providing funds. This study is also being supported by Johns Hopkins University on behalf of the Translational Breast Cancer Research Consortium (TBCRC). The TBCRC is a group of academic medical centers across the United States that work together to conduct breast cancer research.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Participants must have histologically or cytologically confirmed unresectable locally advanced or metastatic invasive breast carcinoma that is HER2-positive by American Society of Clinical Oncology/College of American Pathologists 2018 criteria, as assessed by standard institutional guidelines (central testing is not required). Both estrogen receptor (ER)-positive/HER2-positive and ER-negative/HER2-positive will be eligible.
* Participants with ER-positive disease should continue endocrine therapy.
* Participants must be currently receiving first-line anti-HER2 therapy (any regimen) for metastatic disease and must have been on this therapy for at least 3 years without evidence of progressive disease according to RECIST 1.1 criteria. The following exceptions apply:
* Patients with history of brain-only progressive disease previously treated with local therapy (surgery and/or radiation therapy) are eligible, provided they meet all the following study criteria:

  * Asymptomatic
  * Not requiring anti-convulsant for symptomatic control
  * Not requiring corticosteroids
  * No evidence of interim central nervous system (CNS) progression between the completion of CNS-directed therapy and screening radiographic study
  * Minimum of 2 years (24 months) between completion of CNS-directed therapy and study start
* Participants with history of oligo-progression (i.e., progressive disease of a single lesion) outside CNS treated with local treatment and/or change of endocrine therapy only are eligible, provided they meet the following criteria:

  * No evidence of interval progression between completion of local treatment or endocrine therapy change and screening radiographic study
  * Minimum 2 years (24 months) between completion of local therapy or treatment switch and study start
* CT scan within 30 days of study start without definite evidence of progressive disease in the opinion of the treating investigator.
* Available, representative archival formalin-fixed paraffin-embedded (FFPE) tumor tissue block from primary and/or metastatic site. If tissue block is unavailable, 20 unstained 10uM slides will be accepted (less than 20 slides may be acceptable with documentation of Sponsor-Investigator approval and would not require an eligibility exception). Tumor tissue must be received by coordinating site prior to study enrollment.
* ECOG performance status 0-1
* For intervention arm only (cohort 2): willingness to stop anti-HER2 systemic therapy
* Willingness and ability to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures
* Ability to understand the study requirements and document informed consent indicating awareness of the investigational nature and the risks of this study
* Participants with another prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of this trial are eligible

Exclusion Criteria:

* Participants who are receiving any investigational agents to treat breast cancer
* Participants with psychiatric illness/social situations that would limit compliance with study requirements.
* All English- speaking patients will participate in the PRO measures. Patients that do not read or understand English are eligible to participate but will be exempt from the patient completed questionnaires

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2023-04-19 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2036-02 (Estimated)

PRIMARY OUTCOMES:
1-year progression-free survival (PFS) Stopped Anti-HER2 Treatment | Up to 1 year
  The primary endpoint is one-year progression-free survival (PFS) per RECIST 1.1 assessed separately in the participants who agree to stop HER2 therapy and those who continue HER2 therapy.
1-year progression-free survival (PFS) Continued Anti-HER2 Treatment | Up to 1 year
  The primary endpoint is one-year progression-free survival (PFS) per RECIST 1.1 assessed separately in the participants who agree to stop HER2 therapy and those who continue HER2 therapy.

SECONDARY OUTCOMES:
Clinical benefit rate (CBR) | Up to 1 year
  Determine the clinical benefit rate (CBR) of re-initiation of anti-HER2 therapy for participants who experience disease progression after stopping anti-HER2 therapy. Clinical benefit rate is defined as CR, PR, or SD ≥ 24weeks per RECIST 1.1. Clinical benefit rate after re-initiation of HER2 therapy will be reported with a 95% exact confidence interval.
3-year Overall survival (OS) | Up to 3 years
  Determine 3-year overall survival (OS) in participants in cohorts 1 and 2 using time-to-event analysis methods of Kaplan-Meier
3-year progression-free survival (PFS) | Up to 3 years
  Determine 3-year PFS in participants in cohorts 1 and 2 using time-to-event analysis methods of Kaplan-Meier.
Probability of restarting anti-HER2 Treatment | Up to 1 year
  Proportion of participants that restart anti-HER2 systemic therapy without progression of disease in participants stopping anti-HER2 therapy will be reported with a 95% exact confidence interval.

CONTACTS AND LOCATIONS:
Overall Officials: Nancy U Lin, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (13):
- United States (13):
  - Mayo Clinic Hospital Arizona, Phoenix, Arizona
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - Mayo Clinical Hospital Florida, Jacksonville, Florida
  - Dana-Farber Cancer Insitute, Boston, Massachusetts
  - DFCI @ Foxborough, Foxborough, Massachusetts
  - DFCI @ Merrimack Valley, Methuen, Massachusetts
  - DFCI @ Milford Regional Hospital, Milford, Massachusetts
  - DFCI @ South Shore Hospital, South Weymouth, Massachusetts
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Duke University, Durham, North Carolina
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Baylor College of Medicine, Houston, Texas
  - Fred Hutchinson Cancer Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu
URL: https://www.dana-farber.org/research/innovations